CLINICAL TRIAL: NCT04175600
Title: A Randomized, Multicenter, Double-Blind, Placebo-Controlled, Parallel-Group Study With Open-Label Extension Period to Assess the Efficacy and Safety of Selexipag as Add-On Treatment to Standard of Care in Children Aged >=2 to <18 Years With Pulmonary Arterial Hypertension
Brief Title: A Study of Selexipag as Add-On Treatment to Standard of Care in Children With Pulmonary Arterial Hypertension
Acronym: SALTO
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108716; AC-065A310 (Other: Janssen Research & Development, LLC); 2019-002817-21 (EudraCT Number); 2022-501012-34-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2019-11-08; First posted 2019-11-25 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Hypertension, Pulmonary
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — selexipag

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Selexipag (Experimental): Participants will receive selexipag based on the body weight on Day 1 and will continue thereafter with twice daily dosing. Selexipag will be uptitrated during the first 12 weeks until the participants reaches the individual maximum tolerated dose (iMTD) or until a maximum dose corresponding to their baseline body-weight category is achieved. Uptitration is followed by a maintenance period after Week 12 until end of treatment (EOT), at the maximum tolerated dose.
  Interventions: Drug: Selexipag
- Placebo (Placebo Comparator): Participants will receive matching placebo based on the body weight on Day 1 and will continue thereafter with twice daily dosing.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Selexipag — Selexipag tablet will be administered orally.
  Other Names: JNJ-67896049
  Arms: Selexipag
Drug: Placebo — Matching placebo tablets will be administered orally.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate whether the addition of selexipag to standard of care treatment delays disease progression in children with Pulmonary Arterial Hypertension (PAH) in comparison to placebo.

DETAILED DESCRIPTION:
Pediatric PAH is a rare and progressive disorder associated with considerable morbidity and mortality. Given the significant medical need to develop treatments in children with PAH, further clinical studies in the pediatric population are therefore needed to provide more data for the management of PAH in children. Selexipag (JNJ-67896049) is an orally available, selective, and long-acting non-prostanoid agonist of the prostacyclin receptor approved and commercially available for the treatment of adult participants with PAH. Selexipag and its metabolite possess anti-fibrotic, anti-proliferative, and anti-thrombotic properties. Currently, no medicines targeting prostacyclin pathway are approved for pediatric use in PAH. An effective and orally available therapy acting on the prostacyclin receptor such as selexipag introduced at medically appropriate stage of PAH disease, and primarily in combination with current first-line oral PAH-specific medicines in participants in need of additional therapy because of insufficient disease control would represents a major advance to the therapeutic management of PAH pediatric participants. This study consists of a screening period of up to 6 weeks and a double-blind treatment period, including up-titration and maintenance periods, followed by a 3-year open-label extension period (OLEP) and a 30-day safety follow-up period that occurs after the last dose of study intervention (either double-blind or open-label). Safety, pharmacokinetic and efficacy assessments will be performed during the study. An Independent Data Monitoring Committee (IDMC) will be established to monitor data on an ongoing basis, to review interim data, and to ensure the continuing safety of the participants enrolled in this study. The approximate duration of the study is 8 years.

ELIGIBILITY:
Inclusion Criteria:

* Participants between greater than or equal to (>=) 2 and less than (<) 18 years of age weighing >=9 kilogram (kg) at randomization
* Pulmonary arterial hypertension (PAH) diagnosis confirmed by documented historical right heart catheterization (RHC) performed at any time before participant's screening
* PAH (World Health Organization [WHO] Group 1), including participants with Down syndrome, of the following etiologies: Idiopathic PAH (IPAH); Heritable PAH (HPAH); PAH associated with congenital heart disease (PAH-associated with congenital heart disease [aCHD]) (PAH with coincidental CHD [that is, a small atrial septal defect, ventricular septal defect, or patent ductus arteriosus that does not itself account for the development of elevated PVR] and if approved by the BCAC) and Post-operative PAH (persisting / recurring/ developing >=6 months after repair of CHD); Drug or toxin-induced; PAH associated with Human immunodeficiency virus (HIV)
* WHO functional class (FC) II and III
* Participants treated with at least 1 PAH-specific treatment, example, an Endothelin receptor antagonist (ERA) and/or a Phosphodiesterase type-5 (PDE-5) inhibitor/soluble guanylate cyclase stimulator, provided that the treatment dose(s) has been stable for at least 3 months prior to first dose of study intervention

Exclusion Criteria:

* PAH due to portal hypertension, schistosomiasis, pulmonary veno-occlusive disease, and/or pulmonary capillary hemangiomatosis
* PAH associated with Eisenmenger syndrome
* Previous exposure to Uptravi (selexipag)
* Known concomitant life-threatening disease with a life expectancy <12 months
* Pregnant, planning to become pregnant, or lactating
* Known allergies, hypersensitivity, or intolerance to selexipag or its excipients

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 138 (Actual)
Dates: Start 2020-01-16 (Actual); Primary Completion 2024-10-11 (Actual); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Time to Disease Progression | From randomization up to 7 days after study treatment discontinuation (up to 5 years)
  Time to disease progression is the time from randomization up to 7 days after study treatment discontinuation. Disease progression is defined as the first occurrence of either of the following components: Death (all causes), Atrial septostomy or Potts' anastomosis, or registration on lung transplant list, Hospitalization due to worsening pulmonary arterial hypertension (PAH), Clinical worsening of PAH.

SECONDARY OUTCOMES:
Percentage of Participants with Treatment-emergent Adverse Events (TEAEs) and Serious AEs | Up to 5 years
  An adverse event (AE) is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. TEAEs are AEs with onset during the intervention period or that are a consequence of a pre-existing condition that has worsened since baseline. A SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Percentage of Participants with AEs Leading to Premature Discontinuation of Study Treatment | Up to 5 years
  Percentage of participants with AEs leading to premature discontinuation of study treatment will be reported.
Change from Baseline in Systolic and Diastolic Arterial Blood Pressure | Baseline up to end of treatment (EOT) (up to 8 years)
  Change from baseline in systolic and diastolic arterial blood pressure to all assessed time points will be reported.
Change from Baseline in Pulse Rate | Baseline up to EOT (up to 8 years)
  Change from baseline in pulse rate to all assessed time points will be reported.
Change from Baseline in Body Weight | Baseline up to EOT (up to 8 years)
  Change from baseline in body weight to all assessed time points will be reported.
Change from Baseline in Height | Baseline up to EOT (up to 8 years)
  Change from baseline in height to all assessed time points will be reported.
Sexual Maturation (Tanner Stage) Change from Baseline to all Assessed Time Points | Up to 3 days after study treatment discontinuation (up to EOT) (multiple timepoints up to 8 years)
  The sexual maturation change as per Tanner stage will be assessed from baseline to all assessed time points. Tanner stage I is defined as no pubic hair at all (prepubertal Dominic state); stage II is defined as a small amount of long, downy hair with slight pigmentation at the base of the penis and scrotum (males) or on the labia majora (females); stage III is defined as when the hair becomes more coarse and curly, and begins to extend laterally; stage IV is defined as adult-like hair quality, extending across pubis but sparing medial thighs; and stage V is defined as when the: hair extends to medial surface of the thighs.
Percentage of Participants with Treatment-emergent Electrocardiogram Abnormalities | Baseline up to EOT (up to 8 years)
  Percentage of participants with treatment-emergent electrocardiogram abnormalities will be reported.
Percentage of Participants with Treatment-emergent Marked Laboratory Abnormalities | Baseline up to EOT (up to 8 years)
  Percentage of participants with treatment-emergent marked laboratory (serum chemistry [including pregnancy testing and thyroid markers] and hematology) abnormalities will be reported.
Treatment-emergent Change from Baseline in Thyroid Stimulating Hormone | Baseline up to EOT (up to 8 years)
  Treatment-emergent change from baseline in thyroid stimulating hormone over time will be reported.
Time to First Clinical Event Committee (CEC)-confirmed Hospitalization or Death for PAH | Until 7 days after study treatment discontinuation (Up to 8 years)
  Time to first CEC-confirmed hospitalization or death for PAH is the time (days) from randomization to first occurrence of CEC-confirmed hospitalization for PAH or death due to PAH up to 7 days after study intervention discontinuation.
Trough Plasma Concentration at Steady-state (Ctrough,ss) of Selexipag and its Metabolite ACT-333679 | Weeks 16, 24 and every 12 weeks thereafter (up to 8 years)
  Ctrough,ss is defined as the plasma concentration just prior to the morning dose, with the last study intervention administration one day prior to the pharmacokinetic sampling and will be reported for Selexipag and its metabolite ACT-333679.
Change from Baseline at Week 24 in Log2 N-terminal Pro-brain Natriuretic Peptide (NT-proBNP) | Baseline up to Week 24
  The change from baseline at week 24 in log2 NT-proBNP will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Actelion Clinical Trial, Study Director — Actelion
Locations (114):
- United States (13):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - UCLA Medical Center, Los Angeles, California
  - UCSF, San Francisco, California
  - Childrens Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Congenital Heart Center of the University of Florida, Gainesville, Florida
  - Riley Hospital for Children, Indianapolis, Indiana
  - Detroit Medical Center, Detroit, Michigan
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Childrens Hospital Of Philadelphia, Philadelphia, Pennsylvania
  - Texas Children's Hospital, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Virginia Division of Pediatric Cardiology, Charlottesville, Virginia
- Queensland CHILDREN'S HOSPITAL, South Brisbane, Australia
- Belarus (2):
  - State Institution Republican Scientific And Practical Center For Pediatric Surgery, Minsk
  - Health Institution 4Th City Children'S Clinical Hospital, Minsk
- Belgium (3):
  - ULB Hôpital Erasme, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - Universitaire Ziekenhuizen Leuven, Leuven
- Brazil (8):
  - Complexo de Prevencao,Diagnostico,Terapia e Reabilitacao Respiratoria LTDA Hospital Dia do Pulmao, Blumenau
  - Fundacao Universitaria de Cardiologia - Instituto de Cardiologia e Transplantes do DF, Brasília
  - Hospital Pequeno Principe, Curitiba
  - Secretaria da Saude do Estado do Ceara - Hospital Doutor Carlos Alberto Studart Gomes, Fortaleza
  - Irmandade Santa Casa de Misericordia de Porto Alegre, Porto Alegre
  - Fundacao Universitaria de Cardiologia, Porto Alegre
  - Irmandade Santa Casa de Misericordia de Sao Paulo, São Paulo
  - SPDM - Associacao Paulista para o Desenvolvimento da Medicina - Hospital Sao Paulo, São Paulo
- Multiprofile Hospital For Active Treatment National Cardiology Hospital, Ead, Sofia, Bulgaria
- Canada (2):
  - Stollery Children's Hospital, Edmonton, Alberta
  - Hospital For Sick Children, Toronto, Ontario
- China (6):
  - Beijing Anzhen Hospital, Beijing
  - Guangzhou Women And Children's Medical Center, Guangzhou
  - Qingdao Women and Children's Hospital, Qingdao
  - Shanghai Childrens Medical Center, Shanghai
  - Children's Hospital of Fudan University, Shanghai
  - The General Hospital of Northern Theater Command, Shenyang
- Colombia (6):
  - Clinica San Rafael, Bogotá
  - Fundacion Neumologica Colombiana, Bogotá
  - Fundacion Santa Fe de Bogota, Bogotá
  - Clínica Imbanaco S.A.S., Cali
  - Fundacion Cardiovascular de Colombia, Piedecuesta
  - Hospital Universidad del Norte, Soledad
- New Children's Hospital of the Helsinki University Hospital (HUS), Helsinki, Finland
- France (6):
  - Hôpital Cardiologique - Chru Lille, Lille
  - Hopital de la Timone, Marseille
  - CHU Arnaud de Villeneuve, Montpellier
  - Hôpital Necker - Enfants Malades, Paris
  - Hôpital Cardiologique Du Haut-Lévêque, Pessac
  - Chu Hopital Des Enfants, Toulouse
- Germany (4):
  - Universitätsklinikum Freiburg Zentrum, Freiburg im Breisgau
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Herzzentrum Leipzig GmbH, Leipzig
  - Klinikum der Universitaet Muenchen, München
- Gottsegen György Országos Kardiológiai Intézet, Budapest, Hungary
- Our Lady's Children's Hospital, Dublin, Ireland
- Israel (2):
  - Rambam Medical Center, Haifa
  - Sheba Medical Center, Ramat Gan
- Italy (6):
  - Azienda Ospedaliera Policlinico S. Orsola-Malpighi, Bologna
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Universta Degli Studi Di Padova, Padua
  - Ospedale Pediatrico Bambin Gesù, Roma
  - IRCCS Policlinico San Donato, S. Donato Milanese
  - AOU Città della Salute e della Scienza di Torino, Presidio Ospedale Infantile Regina Margherita, Torino
- Vilnius University Hospital Santariskiu Clinics, Vilnius, Lithuania
- National Heart Institute, Kuala Lumpur, Malaysia
- Mexico (3):
  - CICUM San Miguel, Guadalajara
  - Operadora de Hospitales Angeles SA de CV Hospital Angeles Lomas, México
  - Unidad de Investigacion Clinica en Medicina S.C. (UDICEM), Monterrey
- Poland (6):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Uniwersytecki Szpital Dzieciecy w Krakowie, Krakow
  - Szpital Kliniczny im Karola Jonschera, Poznan
  - Instytut Pomnik Centrum Zdrowia Dziecka, Warsaw
  - Wojewodzki Szpital Specjalistyczny we Wroclawiu, Wroclaw
  - Slaskie Centrum Chorob Serca, Zabrze
- Portugal (2):
  - Uls Sao Jose - Hosp. Santa Marta, Lisbon
  - Uls Sao Joao - Hosp. Sao Joao, Porto
- Russia (5):
  - Kazan State Medical University, Kazan'
  - Cardiovascular Pathology Research Institute of Siberian Branch of RAMS, Kemerovo
  - Childrens City Clinical Hospital n.a. Bashlyaeva, Moscow
  - Veltischev Research and Clinical Institute for Pediatrics of the Pirogov RNRMU, Moscow
  - Samara Regional Clinical Cardiological Dispensary, Samara
- Univerzitetska Dečja Klinika, Belgrade, Serbia
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Pusan National University Yangsan Hospital, Yangsan
- Spain (6):
  - Hosp Univ A Coruna, A Coruña
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp. Sant Joan de Deu, Esplugues de Llobregat
  - Hosp. Gral. Univ. Gregorio Maranon, Madrid
  - Hosp. Univ. La Paz, Madrid
  - Hosp. Virgen Del Rocio, Seville
- Sweden (2):
  - Drottning Silvias barn- och ungdomssjukhus, Gothenburg
  - Skanes universitetssjukhus, Lund
- Centre Hospitalier Universitaire Vaudois CHUV, Lausanne, Switzerland
- Taiwan (3):
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
- Thailand (2):
  - Chiang Mai University Hospital, Chiang Mai
  - Songklanagarind hospital, Songkhla
- Turkey (Türkiye) (6):
  - Cukurova Balcali Hospital Application and Research Center, Adana
  - Hacettepe University Medical Faculty, Ankara
  - CAPA Istanbul University Medical Faculty, Istanbul
  - Mehmet Akif Ersoy Training and Research Hospital, Istanbul
  - Behcet Uz Pediatric Diseases and Surgery Training and Research Hospital, Izmir
  - Izmir Tepecik Training and Research Hospital, Izmir
- Ukraine (4):
  - Dnipropetrovsk clinical medical center of Mother and Child after prof. Rudnev, Dnipro
  - MI 'Dnipropetrovsk Regional Clinical Center of Cardiology and Cardiac Surgery', Dnipro
  - Scientific Practical Medical Center for Pediatric Cardiology and Cardio Surgery of the MOH, Kyiv
  - MI Zaporizhzhia Regional Clinical Childrens Hospital of Zaporizhzhia Regional Council, Zaporizhzhya
- Vietnam (4):
  - Hanoi Medical University Hospital, Hanoi
  - Tam Anh Hospital, Ho Chi Minh City
  - University Medical Center Ho Chi Minh city, Ho Chi Minh City
  - Children's Hospital 1, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency